CLINICAL TRIAL: NCT04449653
Title: Mobile Study to Measure and Predict Lupus Disease Activity Using Digital Signals
Acronym: OASIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Progentec Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MEASURE
Record Dates: First submitted 2020-05-26; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Erythematosus
Keywords: Lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lupus Cases: Individuals who are diagnosed with System Lupus Erythematosus and consent to the study will be placed in this cohort. Upon enrollment they will be given the opportunity to invite a non-SLE-diagnosed friend to enroll in the study as a healthy control. These individuals will answer weekly questions and receive a smartwatch to measure their physical activity.

SUMMARY:
OASIS: A mobile study to measure and predict lupus (SLE) disease activity using digital signals The OASIS study is exploring how patient reported data and digital biomarkers, like activity level and heart rate variability, can be used to predict changes in lupus disease activity. You may receive a Withings Steel HR smartwatch as part of this study. The purpose of this study is to look for factors that affect lupus disease activity and potentially predict lupus flares through non-clinical tests

ELIGIBILITY:
Inclusion Criteria:

* Female or male age 18 or older
* Participant is currently not enrolled in another study
* Able to understand the requirements of the study, provide written informed consent, including consent for the use and disclosure of research-related health information, and comply with the study data collection procedures

Exclusion Criteria:

* NOT able to understand the requirements of the study, provide written informed consent, including consent for the use and disclosure of research-related health information, and comply with the study data collection procedures
* Known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lupus is more common by 3.5-fold among minority groups, e.g., African Americans, than it is among European- Americans.Additionally more than 90% of diagnosed cases of lupus are women. We anticipate significant enrollment of female gender and minority populations reflecting this racial and disparity in disease occurrence rates. Participants will be enrolled from across the United States, with no specific geographic locations being targeted or preferred.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
OASIS Wellness and Disease Questionnaire | Week two
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week three
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week four
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week five
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week six
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week seven
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week eight
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week nine
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week ten
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week eleven
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twelve
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week thirteen
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week fourteen
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week fifteen
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week sixteen
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week seventeen
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week eighteen
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week nineteen
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twenty
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twenty-one
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twenty-two
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twenty-three
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twenty-four
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twenty-five
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
OASIS Wellness and Disease Questionnaire | Week twenty-six
  Basic Health Information and Systemic Lupus Erythematosus-specific questions over the time span of a week
Short Form, 36 question form | Month one
  36 questions asking individuals questions about their general health and wellness, not disease-specific
Short Form, 36 question form | Month two
  36 questions asking individuals questions about their general health and wellness, not disease-specific
Short Form, 36 question form | Month three
  36 questions asking individuals questions about their general health and wellness, not disease-specific
Short Form, 36 question form | Month four
  36 questions asking individuals questions about their general health and wellness, not disease-specific
Short Form, 36 question form | Month five
  36 questions asking individuals questions about their general health and wellness, not disease-specific
Short Form, 36 question form | Month six
  36 questions asking individuals questions about their general health and wellness, not disease-specific
Withings Heartrate & Activity | Continuously, for six months
  Patient activity, sleep quality, and heart rate collected by the wearable watch

SECONDARY OUTCOMES:
Heart rate variability | Week two
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week three
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week four
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week five
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week six
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week seven
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week eight
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week nine
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week ten
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week eleven
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twelve
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week thirteen
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week fourteen
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week fifteen
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week sixteen
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week seventeen
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week eighteen
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week nineteen
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twenty
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twenty-one
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twenty-two
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twenty-three
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twenty-four
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twenty-five
  Measurement of individual's change in pulse via a smartphone's onboard camera
Heart rate variability | Week twenty-six
  Measurement of individual's change in pulse via a smartphone's onboard camera

OTHER OUTCOMES:
OASIS Baseline Questionnaire | Baseline, entered only upon enrollment
  Basic Health Information and SLE-specific questions

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Jupe, Ph.D., Principal Investigator — Progentec Diagnostics
Locations (1):
- Ryan Newhardt, Oklahoma City, Oklahoma, United States